CLINICAL TRIAL: NCT03552146
Title: Evaluation of the Effects on Efficiency of a Sedation Service by Switching From Propofol to Dexmedetomidine
Brief Title: Evaluating the Effects of Propofol vs. Dexmedetomidine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Healthcare of Atlanta (Other)
Collaborators: Morehouse School of Medicine (Other)
Responsible Party: Principal Investigator, David Fagin, MD, Assistant Medical Director, Children's Healthcare of Atlanta
Other Study IDs: 17-136
Record Dates: First submitted 2018-03-30; First posted 2018-06-11 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Sedative Adverse Reaction
Keywords: sedation
MeSH Terms: interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Sedation Group 1: Patients will receive standard of care dose of Propofol, based on the provider's assessment, prior to radiologic procedure.
  Interventions: Drug: Propofol
- Sedation Group 2: Patients will receive standard of care dose of dexmedetomidine, based on the provider's assessment, prior to radiologic procedure.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — Patients will be randomized to either propofol or dexmedetomidine and then observed for sedation-related events from time of drug administration to discharge.
  Other Names: Diprivan
  Groups: Sedation Group 1
Drug: Dexmedetomidine — Patients will be randomized to either propofol or dexmedetomidine and then observed for sedation-related events from time of drug administration to discharge.
  Other Names: Precedex
  Groups: Sedation Group 2

SUMMARY:
The primary purpose of this observational study is to compare what drugs work best in sedating children (> 3 months to < 36 months) who need an MRI. This type of research may help clinicians (healthcare providers) learn more about how dexmedetomidine works compared to propofol. The investigators are planning to have 60 children complete the study at Children's Healthcare of Atlanta at Scottish Rite. Half (30) of the patients will be randomized to receive dexmedetomidine and the other half will receive propofol. (Both drugs are licensed and approved for the sedation performed for consented patients.)

DETAILED DESCRIPTION:
There are several different medications commonly being used to facilitate the administration of radiologic procedures on children. Procedures such as Magnetic Resonance Imaging (MRIs) require that the patient remain still for the duration of the test. Propofol has become the drug of choice for many sedation services due to its rapid onset of action, rapid recovery time, ability to achieve sedation reliably and favorable safety profile. Dexmedetomidine, a selective alpha-2- adrenergic agonist, has also gained popularity with sedation services. Its main advantage over propofol is that it has minimal respiratory complications when compared to propofol. The sedative effect from dexmedetomidine preserves a natural sleep pattern and induces cooperative sedation in which patients are easily arousable. In pediatric studies, the most frequent adverse effect have been related to its potential to cause hypotension and bradycardia, which resolve with dose reduction. Additionally, dexmedetomidine does not seem to have as much impairment of cognitive function and has an opioid sparing effect. Dexmedetomidine, however, has a longer onset of action and longer recovery time compared to propofol, which has limited its use with many sedation services.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (or Parent/Guardian) is English speaking
2. Patient is undergoing a scheduled, elective non-contrast MRI of the brain
3. Patient is > 3 months to <36 months of age

Exclusion Criteria:

1. Patients undergoing MRI with contrast
2. Patients older than 36 months of age or younger than 3 months of age
3. Patients presenting to Emergency Department (ED) out of screening hours
4. Patients who are not English speaking
5. Patients who have history or record of propofol or dexmedetomidine allergy
6. Patients with known or history of anaphylaxis to eggs, egg products, soybeans, or soy based products; if patient has a history of a hypersensitivity reaction associated with exposure to eggs, egg products, soybeans, or soy based products, approval must be given by the treating attending physician and documented on the patient's medical record.
7. Patients with unstable cardiac or respiratory status as determined by treating attending physician
8. Patients who are receiving digoxin

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will draw from children who are scheduled for non emergent sedation to undergo a brain non contrast, magnetic resonance imaging (MRI) study. Children are otherwise healthy and fall within the age span of 3 months to 36 months. This is an observational study of the outcomes outlined, when patients agree to be randomized to either of 2 drugs which are FDA approved to provide optimal sedation for this MRI procedure.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Procedural times to achieve optimal sedation | Start of procedure to discharge (up to 8 hours)
  Measuring the amount of time it takes for a patient to be discharged starting from induction (start of infusion).

SECONDARY OUTCOMES:
Sedation related events | Start of procedure to up to 36 hours post-discharge
  Adverse events related to the sedation (i.e., apnea, desaturation, change in heart rate)

OTHER OUTCOMES:
Post-discharge clinical status | Baseline to 24 hours post discharge
  Recording any events post-discharge that are possibly sedation-related

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a pilot study of observations made of patients who are randomized to receive 1 of 2 sedation medications, which are currently FDA approved for the proposed study. The data will help researchers determine the feasibility to conduct a large scale multi-center study to look specifically at primary outcomes as outlined in the proposal.